CLINICAL TRIAL: NCT03624816
Title: A Randomized, No-treatment Controlled, Evaluator-blinded, Multi-center Study to Evaluate the Effectiveness and Safety of Restylane Defyne in the Chin for Augmentation and Correction of Chin Retrusion
Brief Title: A Study to Evaluate the Safety and Efficacy of Restylane Defyne for Chin Augmentation and Correction of Chin Retrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USCH1702
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Chin Retrusion; Chin Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Restylane Defyne (Experimental): injection with Restylane Defyne
  Interventions: Device: Restylane Defyne
- Control (No Intervention): no-treatment control

INTERVENTIONS:
Device: Restylane Defyne — hyaluronic acid dermal filler gel
  Arms: Restylane Defyne

SUMMARY:
To demonstrate the effectiveness of Restylane Defyne for chin augmentation and correction of chin retrusion by demonstrating the superiority in responder rates relative to no treatment.

DETAILED DESCRIPTION:
This was a randomized, no-treatment-controlled, evaluator-blinded, multi-center study to evaluate the effectiveness and safety of Restylane Defyne in the chin for augmentation and correction of chin retrusion.

This study was designed to enroll and randomize approximately 140 subjects in a 3:1 ratio of treatment to Restylane Defyne or no-treatment-control, including at least 21 subjects of Fitzpatrick skin type IV through VI. All randomized subjects were to have a Galderma Chin Retrusion Scale (GCRS) score of 1 (Mild) or 2 (Moderate).

Eligible subjects randomized to receive treatment were injected by the Treating Investigator at Day 1. The method of injection was at the discretion of the Treating Investigator. A sufficient amount of product was injected to achieve optimal correction of the chin, in the opinion of the Treating Investigator and subject. Optimal appearance was defined as at least 1 GCRS grade improvement from baseline and the best correction that could be achieved as agreed by the Treating Investigator and the subject.

At the 48-week visit, after all study procedures for the visit were completed, treated subjects had the option of receiving an additional treatment if optimal aesthetic improvement was not maintained with Restylane Defyne. Non-treated control subjects also had the option of receiving treatment with Restylane Defyne in the chin at Week 48. If an optional treatment was performed, a safety follow-up visits were scheduled

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to comply with the requirements of the study and providing a signed written informed consent.
* Males or non-pregnant, non-breastfeeding females, 22 years of age or older, seeking chin augmentation or correction of retrusion

Exclusion Criteria:

* Allergy of hypersensitivity to any injectable hyaluronic acid gel or to gram positive bacterial proteins
* Allergy or hypersensitivity to lidocaine or other amide-type anesthetics, or topical anesthetics or nerve blocking agents

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Westside Aesthetics, Los Angeles, California
  - Ablon Skin Institute and Research Center, Manhattan Beach, California
  - Marcus Facial Plastic Surgery, Redondo Beach, California
  - Moradi M.D., Vista, California
  - Skin Research Institute, LLC, Coral Gables, Florida
  - Etre Cometic Dermatology and Laser Center, New Orleans, Louisiana
  - WIDLS Chevy Chase, Chevy Chase, Maryland
  - Maryland Laser Skin and Vein Institute, Hunt Valley, Maryland
  - Union Square Laser Dermatology, New York, New York
  - Wilmington Dermatology and Laser Center, Wilmington, North Carolina
  - Dallas Plastic Surgery Institute, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane Defyne | Control
Started | 107 | 33
Completed | 97 | 26
Not Completed | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restylane Defyne | Control | Total
Number analyzed (Participants) | 107 | 33 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (12.39) | 44.4 (15.30) | 47.4 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 30 | 125
  Male | 12 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 5 | 17
  White | 85 | 22 | 107
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 107 | 33 | 140
Fitzpatrick Skin type (FST) [Count of Participants; unit: Participants] — FST I: white; very fair; red or blond hair; blue eyes; freckles. always burns, never tans.
  FST II: white; fair; red or blond hair; blue, hazel or green eyes. usually burns, tans with difficulty.
  FST III: cream white; fair with any eye or hair color; very common. sometimes mild burn, gradually tans.
  FST IV: brown; typical Mediterranean Caucasian skin. rarely burns, tans with ease.
  FST V: dark brown; Middle Eastern skin types. very rarely burns, tans very easily.
  FST VI: Skin color - black. Skin Characteristics - never burns, tans very easily.
  Participants
    FST I | 7 | 1 | 8
    FST II | 27 | 8 | 35
    FST III | 30 | 10 | 40
    FST IV | 24 | 8 | 32
    FST V | 10 | 4 | 14
    FST VI | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Effectiveness of the Treatment Using the Galderma Chin Restrusion Scale
Description: subjects achieving at least 1-grade improvement from baseline using the Galderma Chin Retrusion Scale (GCRS; 0=no retrusion, 1=mild retrusion, 2=moderate retrusion, 3=substantial retrusion) as assessed by blinded evaluator
Time Frame: 12 weeks after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Defyne | Control
Number analyzed (Participants) | 107 | 33
Participants | 87 | 2

2. Secondary Outcome: Evaluate Subject Satisfaction Using the FACE-Q (Baseline to Week 12)
Description: Summary of change from Baseline to Week 12 in the FACE-Q Satisfaction with Chin, where subjects were asked about their satisfaction with treatment outcome on their chin. Higher scores reflect a better outcome. Scale consists of 10 questions and subjects select level of satisfaction for each question from/to Very dissatisfied = 1, Somewhat dissatisfied = 2, Somewhat satisfied = 3, Very satisfied = 4. A Conversion Table converts raw scale summed score into a score from 0 (worst) to 100 (best). If missing data is less than 50% of the scale's items, the mean of the completed items is used (Rasch Transformed Total Score: BOCF (ITT Population).
Time Frame: 12 weeks after last injection
Population: ITT Population; NOTE: Of the 140 subjects enrolled, 1 subject was randomized but did not complete baseline FACE-Q before withdrawing consent and is, therefore, not included in this table.
Measure: Mean (Standard Deviation); unit: Rasch Transformed Score
Arm/Group | Restylane Defyne | Control
Number analyzed (Participants) | 106 | 33
Rasch Transformed Score | 78.6 (22.14) | 35.1 (21.20)

3. Secondary Outcome: Evaluate Effectiveness of the Treatment Using the Galderma Chin Retrusion
Description: Response rates, defined by at least 1 point improvement from baseline using the Galderma Chin Retrusion Scale (GCRS), as assessed by the Blinded Evaluator, at 24,36, and 48 weeks after the last injection for the treatment group or after baseline if randomized to no treatment
Time Frame: 24, 36, and 48 weeks after last injection
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Defyne | Control
Number analyzed (Participants) | 101 | 31
Participants | 87 | 2

4. Secondary Outcome: Assess Overall Aesthetic Improvement Using the Global Aesthetic Improvement Scale
Description: Aesthetic improvement (overall appearance) after treatment with Restylane® Defyne compared to no-treatment control, as determined by assessments using the Global Aesthetic Improvement Scale (GAIS). Assessments were performed at 12, 24, 36, and 48 weeks after treatment. Treating Investigators and subjects separately rated aesthetic improvement of the chin from baseline appearance, where a higher score reflects reporting of greater improvement. The subjects and Investigators select a score from the following categorical scale: Very much improved = 3; Much improved = 2; Improved = 1; No change = 0; Worse = -1; Much worse = -2; Very much worse = -3. Scores range from -3 (worst) to 3 (best). Higher scores reflect a better outcome. The Responder Rate is defined as the number and percent of subjects with a rating of at least "Improved" based off of subject's/investigator's (as appropriate) assessment of the GAIS.
Time Frame: 12, 24, 36, and 48 weeks after last injection
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Defyne | Control
Number analyzed (Participants) | 101 | 31
Participants | 100 | 0

5. Secondary Outcome: Evaluate Subject Satisfaction Using the FACE-Q (From Baseline to Week 24)
Description: Summary of Change from Baseline to Week 24 in FACE-Q Satisfaction with Chin, where subjects were asked about their satisfaction with treatment outcome on their chin. Higher scores reflect a better outcome. Scale consists of 10 questions and subjects select level of satisfaction for each question from/to Very dissatisfied = 1, Somewhat dissatisfied = 2, Somewhat satisfied = 3, Very satisfied = 4. A Conversion Table converts raw scale summed score into a score from 0 (worst) to 100 (best). IIf missing data is less than 50% of the scale's items, the mean of the completed items is used (Rasch Transformed Total Score: BOCF (ITT Population).
Time Frame: 24, 36, and 48 weeks after last injection
Population: ITT population
Measure: Mean (Standard Deviation); unit: FACE-Q Satisfaction with Chin Rasch Tran
Arm/Group | Restylane Defyne | Control
Number analyzed (Participants) | 98 | 30
FACE-Q Satisfaction with Chin Rasch Tran | 75.9 (21.76) | 33.2 (20.77)

6. Secondary Outcome: Evaluate Volume Change in the Treated Area Using 3D Imaging
Description: Summary of Total Volume Change in the Chin Area Measured by Digital 3D Photography at Each Visit (ITT Population). Total volume change corresponds to net volume change from baseline in the chin area.
Time Frame: 12, 24, 36, and 48 weeks after last injection
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Restylane Defyne | Control
Number analyzed (Participants) | 101 | 31
mL
  Week 12 | 3.0 (2.61) | -0.6 (1.46)
  Week 24 | 2.5 (2.34) | -0.3 (1.5)
  Week 36 | 2.5 (2.61) | -0.5 (1.45)
  Week 48 | 2.6 (2.51) | -0.5 (1.14)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Groups:
- Control: Subjects randomized to no treatment/control at baseline
- Restylane Defyne: Subjects randomized to treatment with Restylane Defyne at baseline
  Restylane Defyne: hyaluronic acid dermal filler gel
Arm/Group | Control | Restylane Defyne
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/107
Other Adverse Events (participants affected / at risk) | 10/33 | 65/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=33) | Restylane Defyne (N=107)
Stage IV metastatic lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=33) | Restylane Defyne (N=107)
Implant site pain (General disorders) | 1 (1) | 5 (7)
Implant site bruising (General disorders) | 0 (0) | 3 (3)
Implant site swelling (General disorders) | 0 (0) | 3 (3)
Implant site erythema (General disorders) | 0 (0) | 2 (2)
Implant site hemorrhage (General disorders) | 0 (0) | 2 (2)
Implant site nodule (General disorders) | 1 (1) | 1 (2)
Implant site mass (General disorders) | 0 (0) | 1 (1)
Implant site oedema (General disorders) | 0 (0) | 1 (1)
Implant site eczema (General disorders) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
fatigue (General disorders) | 0 (0) | 1 (1)
implant site cyst (General disorders) | 0 (0) | 1 (1)
influenza like illness (General disorders) | 0 (0) | 1 (1)
injection site eczema (General disorders) | 0 (0) | 1 (1)
nodule (General disorders) | 0 (0) | 1 (1)
pain (General disorders) | 0 (0) | 1 (1)
pyrexia (General disorders) | 0 (0) | 1 (1)
cystitis (Infections and infestations) | 0 (0) | 1 (1)
gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 0 (0) | 1 (1)
tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
oral herpes (Infections and infestations) | 0 (0) | 1 (1)
tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0)
sinusitis (Infections and infestations) | 1 (1) | 0 (0)
contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
procedural anxiety (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
metastases to CNS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1)
presyncope (Nervous system disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 1 (1)
glaucoma (Eye disorders) | 1 (1) | 0 (0)
hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1)
food allergy (Immune system disorders) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree not to present or publish any data or reports collected individually or by subgroup of sites prior to full, initial publication based on all data obtained from all sites.

DOCUMENTS (2):
  • Study Protocol (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT03624816/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT03624816/SAP_001.pdf